CLINICAL TRIAL: NCT01152944
Title: Mechanisms of Stroke in Intracranial Stenosis and Stenting
Brief Title: Mechanisms of Stroke in Intracranial Stenosis
Acronym: MoSIS
Status: Terminated | Type: Observational
Why Stopped: The affiliated study SAMMPRIS (Stenting and Aggressive Medical Management for Preventing Recurrent stroke in Intracranial Stenosis) has stopped enrollment.
Sponsor: Jose Romano, MD (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Jose Romano, MD, Associate Professor of Neurology. Director of Cerebrovascular Division, University of Miami
Organization: University of Miami (Other)
Other Study IDs: 1R01NS069938-01 (NIH); 1R01NS069938-01 (NIH)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Stroke
Keywords: Symptomatic intracranial atherosclerotic disease enrolled in the medical arm of SAMMPRIS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this SAMMPRIS-affiliated study is to understand the mechanisms the mechanisms that underlie ischemic stroke recurrence in high-grade intracranial atherosclerotic disease in order to determine predictors of recurrent stroke. MoSIS will evaluate 6 specific mechanisms of stroke in the medically-treated SAMMPRIS cohort: decreased antegrade flow, progression of stenosis, decreased proximal collateral flow, decreased distal collateral flow, impaired cerebrovascular reserve, and artery-to-artery embolism.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the medical arm of SAMMPRIS, signed consent

Exclusion Criteria:

* For QMRA testing: contraindications to MRI; for TCD testing, abscence of ultrasonographic windows.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical arm of the SAMMPRIS trial which includes recently symptomatic (<30 days) high grade (70% or more)intracranial stenosis of the carotid, middle cerebral, vertebral or basilar arteries.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Ischemic stroke in the territory of the stenotic artery | 2 years from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States